CLINICAL TRIAL: NCT05066633
Title: The Efficacy and Safety of Metoprolol as add-on Treatment to Standard of Care in Preventing Cardiomyopathy in Patients With Duchenne Muscular Dystrophy Aged 8-16 Years. A Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Efficacy and Safety of Metoprolol as add-on Treatment to Standard of Care in Preventing Cardiomyopathy in Patients With DMD
Acronym: MeDMD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBK 154/1/2020; 2020-004901-29 (EudraCT Number)
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Matching placebo will be supplied by the sponsor in child-proof bottles containing dividable tablets with the following dosage of 25mg of IMP and 100mg of IMP. The drug will be administered orally at singular daily doses ranging from 0.75 to 4.5 mg/kg over a Double-Blind Treatment Period (DBTP) of up to 60 months or less dependently on the time of enrolment. The Treatment Period will begin with up to 12-weeks long Up-titration Phase, during which the dose will be gradually escalated. If patient presents with signs and symptoms of intolerance the dose may be temporarily or permanently downgraded at the discretion of the clinician. The up titration ends with reaching maximal tolerated dose level or at a dose corresponding to 4.5 mg/kg.
  Interventions: Drug: Placebo
- Treatment Group (Experimental): Metoprolol succinate will be supplied by the sponsor in child-proof bottles containing dividable tablets with the following dosage of 25mg of IMP and 100mg of IMP. The drug will be administered orally at singular daily doses ranging from 0.75 to 4.5 mg/kg over a Double-Blind Treatment Period (DBTP) of up to 60 months or less dependently on the time of enrolment. The Treatment Period will begin with up to 12-weeks long Up-titration Phase, during which the dose will be gradually escalated. If patient presents with signs and symptoms of intolerance the dose may be temporarily or permanently downgraded at the discretion of the clinician. The up titration ends with reaching maximal tolerated dose level or at a dose corresponding to 4.5 mg/kg.
  Interventions: Drug: Metoprolol Succinate

INTERVENTIONS:
Drug: Metoprolol Succinate — Metoprolol Succinate will be in the form of tablets and will be administered orally once daily. The dose will depend on the patient's weight category. Subject should take their treatment at a consistent time each day to promote compliance. IMP will be up titrated. Every two weeks the patients will be given the higher dose of metoprolol succinate or placebo accordingly to scheme.
  Arms: Treatment Group
Drug: Placebo — Placebo will be in the form of identical tablets and will be administered orally once daily.
  Arms: Control Group

SUMMARY:
The study includes 150 patients with DMD diagnosis confirmed by genetic testing, 8-16 years old (≥8 and <17) at the study entry with a follow-up of up to 5 years. Random enrollment of a patient to one of two groups (intervention or control) takes place after pre-screening and screening stage starts the first phase of the trial. To be eligible for participation in the study, patients must receive standard of care cardiac therapy, which is an Angiotensin-converting-enzyme inhibitor (ACEi) for at least one-month prior to enrollment. A major part of the trial is equal for all patients - who will be receiving indistinguishable investigational medicinal products (IMPs), the drug metoprolol succinate or placebo. As a part of the clinical trial, diagnostic examinations evaluating progression of the disease, will be performed periodically. In addition, all patients will be monitored at home. Heart rate, blood pressure and patients' personal well-being will be controlled using telemedicine technologies. Additional visits in the research center will be provided if any adverse events occur. This model will be continued for 30 months from the enrollment of a first patient. After this period the first drug efficiency analysis will be performed. After that, the intervention may be continued or in case of negative impact of the intervention on patients' health and well-being, terminated with further patients monitoring.

DETAILED DESCRIPTION:
Patients will be evaluated for inclusion during a Screening period of up to one year (possible to extend for another year if warranted). Written informed consent from the patient and/or parent/legal guardian and assent, if applicable, to participate in the study must be obtained prior to beginning any study-related procedures. Once eligibility is confirmed, patients will undergo Screening Assessments.

Two groups will receive either metoprolol succinate (Treatment 1 - Intervention) at a dose depending on the weight category as described below or matching placebo (Treatment 2 - Control) to maintain the study blinding, one per day for up to 60 months. All patients (both arms) will receive ACEi (e.g. perindopril, enarenal, lisinopril) or, if indicated, ARB (e.g. losartan) as a standard of care at an appropriate therapeutic dose (see below) through all the study duration. A total of approximately 150 subjects will be randomized into the study.

Subjects will be assessed for safety and tolerability, clinical efficacy, at scheduled visits throughout the study. Adverse events, including SAEs, and concomitant medications will be recorded throughout the study in eCRF record.

Access credentials for ePROP will be dispensed to the participant or his legal guardian when appropriate at the Enrolment Visit to record vital signs (HR and NIBP) and peak-flow-meter readings, AEs, changes to concomitant medications taken during the study, and any missed or incomplete doses of study medication.

Site study staff will contact the parent(s)/ legal guardian(s) by telephone at quarterly to ensure that the tablet dispensing is proceeding according to protocol and to address any questions the parent(s)/guardian(s) may have.

All subjects will periodically return to the clinical site for assessments according to the Visit Plan. The study is comprised of a Pre-screening, Screening-Enrolment-Randomization Double-Blind Treatment Period further subdivided into Phases.

Subjects will be enrolled into this study at the time written informed consent is given and randomized to treatment only after completion of all Pre-treatment Screening and Enrolment assessments.

Study drug dosing will occur at home on all days starting from Enrolment Visit until the Final Visit.

In the event that relevant clinical or laboratory parameters remain abnormal at the time of discharge from the study, the subject will be followed medically, as clinically indicated.

Any subject who prematurely discontinues the study should return to the study centre for scheduled assessments at the time of early withdrawal, whenever possible assuming the subject has not withdrawn consent.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent(s) or legal guardian(s) has (have) provided written informed consent, where applicable, prior to any study-related procedures; participants will be asked to give written or verbal assent according to requirements (>16 years old)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Ability to take oral medication and be willing to adhere to the study intervention regimen
* Subject has confirmed diagnosis of DMD, as defined as clinical picture consistent with typical DMD and: i) Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, or ii) Identifiable mutation within the DMD gene (deletion/duplication of one or more exons), where reading frame can be predicted as 'out-of-frame' or, iii) Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, other) that is expected to preclude production of the dystrophin protein (i.e., nonsense mutation, deletion/duplication leading to a downstream stop codon)
* Taking ACEi treatment at minimum required doses for at least 30 days

Exclusion Criteria:

* Current or previous permanent use of any beta-blocker medication
* Treatment with another investigational drug or other intervention within 3 months prior to screening
* Clinically significant bradycardia at rest or by Holter ECG, based on age and sex adjusted normal values, atrioventricular block higher than first degree at rest, or second degree Wenckebach at night, pauses longer than 2.5 seconds
* Presence of pacemaker or ICD
* Clinical signs or symptoms of heart failure
* Left ventricular Ejection Fraction (LVEF) <57% (assessed by Teichholtz echocardiography)
* Inability to obtain adequate quality echocardiography images (necessary to monitor for primary endpoint and safety)
* Known allergic reactions to components of the IMPs

Ages: 8 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF %) by Teichholtz method (echocardiography), compared to baseline at Interim Analysis and Final Analysis. | 24 months
  To evaluate whether metoprolol succinate in addition to standard of care treatment compared to placebo in children with DMD delays the progression of LV function loss.

SECONDARY OUTCOMES:
DFS (the time to develop clinically evident heart failure) | 24 months
  To evaluate whether metoprolol succinate in addition to standard of care treatment compared to placebo in children with DMD delays progression of cardiomyopathy and heart failure
Prevalence of patients with myocardial fibrosis assessed by LGE Cardiac magnetic resonance (CMR) | 24 months
  To evaluate whether metoprolol succinate in addition to standard of care treatment compared to placebo in children with DMD delays progression of LGE in CMR
Prevalence of patients with sinus tachycardia based on resting HR (ECG) or defined as mean daily heart rate above 95th percentile for age and sex | 24 months
  To evaluate whether metoprolol succinate in addition to standard of care treatment compared to placebo in children with DMD prevents sinus tachycardia commonly seen in DMD patients
The rate of AE and SAE | 24 months
  To assess the safety and tolerability of metoprolol succinate in children with DMD

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Centre in Gdańsk, Clinic of Paediatric Cardiology and Congenital Heart Defects, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official website — https://medmd.gumed.edu.pl/